CLINICAL TRIAL: NCT01398709
Title: Study of the Relationship Between Rewarming Rate During Cardiopulmonary Bypass and Clinical Prognosis in Infants Undergoing Cardiac Surgery
Brief Title: Effect of Rewarming Rate During Cardiopulmonary Bypass on Clinical Prognosis of Infants Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Chunhu Gu, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Guch-011
Record Dates: First submitted 2011-07-11; First posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; Rewarming Rate
Keywords: Cardiopulmonary Bypass; Prognosis; Cardiac Surgery; Rewarming Rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Slow rewarming strategy (Active Comparator): Slow rewarming strategy (0.24 degrees C/min)
  Interventions: Other: Slow rewarming strategy
- Fast rewarming strategy (Active Comparator): Fast rewarming strategy (0.5 degrees C/min)
  Interventions: Other: Fast rewarming strategy

INTERVENTIONS:
Other: Slow rewarming strategy — Rewarming rate:0.24 degrees C/min.
  Arms: Slow rewarming strategy
Other: Fast rewarming strategy — Rewarming rate:0.5 degrees C/min.
  Arms: Fast rewarming strategy

SUMMARY:
The purpose of this study is to investigate the relationship between rewarming rate during cardiopulmonary bypass and clinical prognosis in infants undergoing cardiac surgery.

DETAILED DESCRIPTION:
There have been many studies indicating that rewarming management plays an important role in cardiac surgery. The purpose of this study is to investigate the relationship between rewarming rate during cardiopulmonary bypass and clinical prognosis in patients undergoing cardiac surgery. Infants undergoing cardiac surgery with cardiopulmonary bypass are randomly assigned to either a slow rewarming strategy (0.24 degrees C/min) or a fast rewarming strategy (0.5 degrees C/min).

ELIGIBILITY:
Inclusion Criteria:

* Infants who had underwent cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Preoperative liver or kidney disease or dysfunction
* Preoperative coagulation disorder
* Palliative operation or a second operation
* Above 3 years

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

SECONDARY OUTCOMES:
Acute renal failure | one month
Respiratory failure | one month
ICU and hospital length of stay, and ICU readmissions | one month
Stroke and reversible ischemic neurologic deficit | one month
Measures of inflammation | one month
  Measures of inflammation (C-reactive protein, TNF-alpha; IL-6) and oxidative stress markers
Biochemical markers of myocardial necrosis | one month
  Biochemical markers of myocardial necrosis（troponin and creatine kinase MB）
Perioperative complications | one month
  Perioperative complications include sternal wound infection (deep and superficial), bacteremia, pneumonia, and major cardiovascular events (acute myocardial infarction, congestive heart failure, and cardiac arrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Dinghua Yi, MD, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China